CLINICAL TRIAL: NCT07201155
Title: The Accuracy of Continuous Glucose Monitoring Systems in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-052
Record Dates: First submitted 2025-06-24; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hyperglycemia in Critically Ill Patients
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Continuous Glucose Monitoring Systems — A trained research member placed the AiDEX® Dynamic Continuous Glucose Monitoring System (Microtech Medical Devices (Hangzhou) Co., Ltd.) on the patient's abdomen, about 3-10 cm to the left or right of the navel, or on the back of the upper arm, according to the instructions. The sensor began to collect data 1-4 hours after successful activation, recording blood glucose values every 5 minutes for 7 consecutive days. For patients who stayed in the ICU for less than 7 days, the continuous glucose monitoring (CGM) was terminated on the day of ICU discharge, and the CGM device was removed.
  Patients monitored their blood glucose using fingerstick point-of-care (POC) measurements every 1-6 hours as needed and had routine arterial blood gas analysis 4-6 times a day. After 24 hours of patient wear, the arterial blood gas glucose (aBG) was used to calibrate the CGMS device at least twice a day. Nurses recorded CGMS data paired with POC values and aBG values in a 1:1 format.
Device: Continuous Glucose Monitoring — This study is a single-center, prospective, observational study conducted in the Intensive Care Unit (ICU) of Nanfang Hospital, Southern Medical University, from May 2024 to August 2024. Patients with elevated blood glucose levels (BG>180 mg/dL) undergoing intravenous insulin therapy were included. Simultaneous blood glucose monitoring was performed using fingerstick blood samples and arterial blood gas analysis, along with the installation of CGMS for concurrent monitoring. CGMS data (CGM values) were recorded in a 1:1 paired format with fingerstick point-of-care (POC) values and arterial blood gas (aBG) values. The correlation of paired blood glucose data was examined using Pearson's correlation coefficient. The accuracy of CGMS was assessed using metrics such as Mean Absolute Relative Difference (MARD), ISO 15197-2013, CLSI POCT12-A3, and Clarke Error Grid Analysis, analyzed with R v.4.4.1 software.
Device: Continuous Glucose Monitoring — Patients who met the inclusion and exclusion criteria were enrolled in the study after obtaining informed consent from the patient or their legal representative. A trained research member placed the AiDEX® Dynamic Continuous Glucose Monitoring System (Microtech Medical Devices (Hangzhou) Co., Ltd.) on the patient's abdomen, about 3-10 cm to the left or right of the navel, or on the back of the upper arm, according to the instructions. The sensor began to collect data 1-4 hours after successful activation, recording blood glucose values every 5 minutes for 7 consecutive days. For patients who stayed in the ICU for less than 7 days, the continuous glucose monitoring (CGM) was terminated on the day of ICU discharge, and the CGM device was removed.
Device: CGMS — Patients who met the inclusion and exclusion criteria were enrolled in the study after obtaining informed consent from the patient or their legal representative. A trained research member placed the AiDEX® Dynamic Continuous Glucose Monitoring System (Microtech Medical Devices (Hangzhou) Co., Ltd.) on the patient's abdomen, about 3-10 cm to the left or right of the navel, or on the back of the upper arm, according to the instructions. The sensor began to collect data 1-4 hours after successful activation, recording blood glucose values every 5 minutes for 7 consecutive days. For patients who stayed in the ICU for less than 7 days, the continuous glucose monitoring (CGM) was terminated on the day of ICU discharge, and the CGM device was removed.

SUMMARY:
Abstract: Hyperglycemia, hypoglycemia, and glucose variability in ICU patients are associated with adverse outcomes. Continuous Glucose Monitoring Systems (CGMS) offer dynamic glucose monitoring and early warnings to improve glucose management. This study aims to evaluate the accuracy and reliability of the CGMS (Microtech AiDEX®) in critically ill patients and its performance under acidosis conditions, providing evidence for its application in the ICU.

Methods: This prospective observational study included patients with BG>180 mg/dL on intravenous insulin therapy. Blood glucose was monitored using point-of-care (POC), arterial blood gas analysis (aBG), and CGMS. CGMS values were paired 1:1 with POC and aBG values. CGMS accuracy was evaluated using MARD, ISO 15197-2013, CLSI POCT12-A3, and Clarke Error Grid Analysis.

ELIGIBILITY:
Inclusion criteria included

1. Age ≥18 years and ≤75 years;
2. Expected ICU stay of at least 3 days;
3. Elevated blood glucose (BG >180 mg/dL) requiring intravenous insulin therapy;
4. Informed consent obtained from the patient or their legally authorized representative.

Exclusion criteria included

1. Severe hepatic failure (Child-Pugh class C) or marked liver dysfunction (total bilirubin ≥50 μmol/L and alanine aminotransferase ≥3 times the upper limit of normal);
2. Uncorrected diabetic ketoacidosis; ability to self-feed; planned magnetic resonance imaging (MRI) examination;
3. Pregnancy or breastfeeding;
4. Extensive skin burns, dermatitis, or severe infections precluding the use of a continuous glucose monitoring system;
5. Severe brain injury, brain death, or moribund state;
6. Deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: blood glucose (BG>180 mg/dL) undergoing intravenous insulin therapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
MARD | From enrollment to discharge/completion of 14-day CGMS wear.
  MARD was calculated as the average of absolute percentage differences between paired glucose measurements: MARD = (1/n) × Σ(|CGMS-Reference|/Reference) × 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China